CLINICAL TRIAL: NCT04809727
Title: Histopathological Findings in Symptomatizing Patients After Supracervical Hysterectomy
Acronym: HSTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Assistant professor, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HistopathSTH
Record Dates: First submitted 2021-03-13; First posted 2021-03-22 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: CIN; Cancer of Cervix; Cervicitis
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervicitis

STUDY DESIGN:
Intervention Model Description: All patients suffering after supracervical hysterectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy (Experimental): four quadrant biopsy
  Interventions: Procedure: Cervical biopsy

INTERVENTIONS:
Procedure: Cervical biopsy — 4 quadrant biopsy

SUMMARY:
Supracervical hysterectomy is widely common and had many complications either immediate or delayed. In these patients bleeding, infection, chronic pelvic pain are common. In these patients cervical biopsy was done and histopathological examinations were done to evaluate the pathology in these patients.

DETAILED DESCRIPTION:
* Study design and settings: Cross sectional descriptive studies conducted from December 2017 till January 2021.
* Patients: 80 patients with supracervical hysterectomy recruited at Tanta University Hospital, gynecology clinics will be recruited according inclusion and exclusion criteria. Inclusion criteria include all symptomatizing patients following supracervical hysterectomy, of any age, of any complaints. The exclusion criteria were patients with total hysterectomy, hysterectomies for malignant indications, and refusal to participate.
* Methods: All patients' demographic data, history, indication of hysterectomy, duration since operation, postoperative complications and their main complaint.

Intervention: under general anesthesia cervical biopsy (4 quadrants) were taken from all patients and was sent for histopathological examinations.

ELIGIBILITY:
Inclusion Criteria:

* all symptomatizing patients following supracervical hysterectomy,

Exclusion Criteria:

* with total hysterectomy,
* hysterectomies for malignant indications,
* refusal to participate.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Detection of cervical neoplasia or cancer incidence | 1 year
  Detection of number of cases diagnosed with cervical Cervical intraepithelial neoplasia, or malignancy by histopathological examination
Detection of chronic cervicitis incidence | 1 year
  Detection of number of cases diagnosed with inflammatory cells and other markers of inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Ayman Shehata Dawood, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided